CLINICAL TRIAL: NCT06624501
Title: Integrated Discovery and Development of Innovative TB Diagnostics
Acronym: (CETR)
Status: Completed | Type: Observational
Sponsor: Harvard University Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Molly Franke, Assistant Professor of Global Health and Social Medicine, Harvard University Faculty of Medicine
Other Study IDs: 5U19AI109755-04 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2020-08

CONDITIONS: Tuberculosis, Pulmonary
Keywords: pediatric; diagnostic; cell-free DNA; molecular; tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Disease; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study maintains a biobank of 9 different sample types collected from children and adults, including: nasopharyngeal swabs, oral swabs, urine, stool, gastric aspirates, sputum, plasma and whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children and adults: Children with symptoms of TB and adults with smear-positive or smear-negative pulmonary TB.
  Interventions: Other: Observational cohort study

INTERVENTIONS:
Other: Observational cohort study

SUMMARY:
The long term goal of this project is to provide information critical to the development and use of a low-cost, point-of-care, rapid, simple, and highly accurate diagnostic tool that can help clinicians make a microbiological diagnosis in children who present with signs and symptoms suggestive of TB.

Specific aim 1: To identify the types of patient samples from which to best detect Mtb DNA in children with TB. We propose to obtain serial samples of sputum, blood, stool, and gastric and nasopharyngeal secretions from children with symptomatic TB and to use molecular methods to characterize the distribution of Mtb in these samples. The results of this study will allow us to identify the most promising sampling strategies for diagnosis of TB in children so that optimization of these easily-accessible samples for detection of Mtb nucleic acids can be addressed.

Specific aim 2: To determine whether cell free Mtb DNA can be detected in plasma and urine samples of children and adults with TB and to describe the host-related factors that alter the sensitivity of this assay. We propose to test serial urine and plasma samples for Mtb DNA fragments in two groups: (1) children with symptoms of TB and (2) adults with TB. Here, we will optimize sample volume sizes and of state-of-the-art sequencing tools to improve DNA recovery and detection. This study will help identify optimal samples and strategies for the non-invasive diagnosis of Mtb using urine.

Secondary aim: To create a bank of archived specimens for (1) optimization of Mtb DNA purification, extraction, and (2) use in future pediatric TB diagnostic research.

ELIGIBILITY:
Inclusion Criteria for aim 1:

Children must meet all of the following criteria at the time of enrollment to participate:

* Age < 15 years;
* Presents to a participating health center;
* Meets the Criteria for Enrollment of Children Into TB Diagnostic Evaluation Studies
* Has a history of contact with an adult with TB disease; and
* A guardian provides informed consent for minor to participate and, if age 8 to 14 years, the minor also provides assent.

Inclusion criteria for aim 2:

Inclusion criteria for children who participate in Aim 2 will be the same as for those for Aim 1. Adults who participate in Aim 2 must meet all of the following criteria at the time of enrollment to participate.

* Age ≥ 18 years;
* Presents to a participating health center;
* Is diagnosed with incident pulmonary TB;
* Has sputum smear microscopy results;
* Has not yet initiated tuberculosis treatment; and
* Is willing to receive a rapid HIV test.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise (1) children (0-14 years) with symptoms of tuberculosis disease (TB) and (2) adults >18 years of age with a diagnosis TB. All participants will be recruited from Lima, Peru.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity for detection of Mtb, by sample type | Baseline
  For each type of biologic specimen, the proportion of samples in which Mtb could be isolated by DNA detection methods (sensitivity) relative to the standard of care (a combination of sputum smear, sputum culture, signs and symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Molly F. Franke, ScD, Principal Investigator — Harvard Medical School (HMS and HSDM)

IPD SHARING:
Plan to Share IPD: No